CLINICAL TRIAL: NCT05799833
Title: The Prevalence and Significance of Low QRS Voltages in Young Healthy Individuals and Athletes
Brief Title: Low QRS Voltages in Young Healthy Individuals and Athletes
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Imperial College London (Other)
Collaborators: Royal Brompton & Harefield NHS Foundation Trust (Other); Cardiac Risk in the Young (Other); St George's, University of London (Other)
Responsible Party: Sponsor
Other Study IDs: 22IC7985; WHCC_PA2965 (Other Grant/Funding Number: Royal Brompton Hospital charity)
Record Dates: First submitted 2023-03-23; First posted 2023-04-05 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-10

CONDITIONS: Sudden Cardiac Death; Sudden Cardiac Arrest; Sudden Cardiac Death Due to Cardiac Arrhythmia; Arrhythmogenic Right Ventricular Cardiomyopathy; Arrhythmogenic Left Ventricular Cardiomyopathy; Dilated Cardiomyopathy
Keywords: Low QRS Voltage; Low QRS amplitude; Sudden Cardiac Death; Cardiac magnetic resonance; Myocardial fibrosis; Premature Ventricular complexes; Dilated Cardiomyopathy; Arrythmogenic right ventricular cardiomyopathy; Arrhythmogenic Left Ventricular Cardiomyopathy; Late Gadolinium Enhancement; Implantable cardioverter defibrillator; Cardiopulmonary exercise testing; Athletes; Genetic inheritance; Non sustained ventricular tachycardia; Pre participation screening; Sports screening
MeSH Terms: conditions — Death, Sudden, Cardiac; Arrhythmogenic Right Ventricular Dysplasia; Cardiomyopathy, Dilated; Ventricular Premature Complexes | interventions — Hematologic Tests; Genetic Testing

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples obtained from each participant for the purpose of performing genetic testing to identify protein altering genetic variants in known genes associated with ARVC/DCM.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Athletes with low QRS voltage: Cohort (anticipated N = 60) will undergo testing with 12 lead ECG, blood test, cardiac MRI, 24 hour holter monitoring and cardiopulmonary exercise testing.
  A subgroup of those identified to have low QRS voltage and myocardial scar on CMR will undergo genetic testing (anticipated number to be tested, N= 25)
  Interventions: Diagnostic Test: Cardiovascular magnetic resonance scan - 3T scanner (Siemens Vida)
- Young healthy individuals (non-athletes) with low QRS voltage: Cohort (anticipated N = 60) will undergo testing with 12 lead ECG, blood test, cardiac MRI, 24 hour holter monitoring and cardiopulmonary exercise testing.
  A subgroup of those identified to have low QRS voltage and myocardial scar on CMR will undergo genetic testing (anticipated number to be tested, N= 25)
  Interventions: Diagnostic Test: Cardiovascular magnetic resonance scan - 3T scanner (Siemens Vida)
- Age and sex matched control group of athletes with normal QRS voltage: Cohort (anticipated N = 60) will undergo testing with 12 lead ECG, blood test, cardiac MRI, 24 hour holter monitoring and cardiopulmonary exercise testing.
  Interventions: Diagnostic Test: Cardiovascular magnetic resonance scan - 3T scanner (Siemens Vida)
- Age and sex matched young healthy controls (non-athletes) with normal QRS voltage: Cohort (anticipated N = 60) will undergo testing with 12 lead ECG, blood test, cardiac MRI, 24 hour holter monitoring and cardiopulmonary exercise testing.
  Interventions: Diagnostic Test: Cardiovascular magnetic resonance scan - 3T scanner (Siemens Vida)

INTERVENTIONS:
Diagnostic Test: Cardiovascular magnetic resonance scan - 3T scanner (Siemens Vida) — 4 study groups will undergo testing with 12-lead ECG, blood test, cardiac MRI, cardiopulmonary exercise testing and 24 hour holter monitor. A subgroup (N=50 anticipated) will undergo genetic testing.
  Other Names: Cardiopulmonary exercise test - COSMED E100w upright cycle ergometer; 24 hour holter monitor - Lifecard CF Holters; Blood test for thyroid function and genetic testing (whole exome sequencing on the Illumina sequencing platform)

SUMMARY:
There is some limited evidence that reduced size of electrical complexes/traces of the heart on the electrocardiogram (ECG) may be associated with scarring in the heart muscle, which may predispose to serious life-threatening electrical abnormalities and sudden cardiac death (SCD). There is no current guidance on how young individuals and athletes with reduced ECG traces should be managed. Therefore, correct interpretation of this ECG finding is crucial for identifying athletes with disease and at risk of SCD. Some athletes experience SCD despite normal standard cardiac tests. The investigators, therefore, propose to study young healthy individuals and young athletes using cardiovascular MRI, cardiopulmonary exercise testing, 24 hour ECG monitoring and genetic analysis to determine the significance of reduced ECG traces and possibly revise current international sports recommendations.

DETAILED DESCRIPTION:
There is emerging evidence that low QRS voltages <0.5mV in the limb leads may be associated with left ventricular myocardial fibrosis and a predisposition to serious ventricular arrhythmias and sudden cardiac death (SCD). Sudden death in young individuals is highlighted most commonly when an athlete is affected. A proportion of decedents are diagnosed with idiopathic myocardial fibrosis at autopsy. Recent studies have revealed myocardial fibrosis in athletes with low QRS complexes, who have survived a sudden cardiac arrest. Low QRS voltages do not feature in the electrical anomalies that warrant further investigation according to the international recommendations for electrocardiographic (ECG) interpretation in athletes, hence there is no information on the precise significance or outcome data in athletes with small QRS voltages. The investigators postulate that further evaluation of athletes with low QRS voltages using CMR and gene analysis will help determine the prevalence and significance of these ECG changes potentially identifying young vulnerable individuals at risk of SCD. There are currently 2 studies which have assessed small QRS complexes in athletes. These studies revealed 1.1-4% of Italian athletes had small QRS complexes. One study performed ultrasound of the heart showing that athletes in general had larger hearts compared to sedentary counterparts but no evidence of structural disease. The second study did not perform CMR in all athletes with small QRS complexes and only conducted CMR in 5 athletes with small QRS complexes and electrical issues and demonstrated scar in 2 athletes. The scientific basis of these studies does not prove the precise significance of small QRS complexes on the ECG in this population to elucidate the sensitivity and specificity of disease identification. It is possible that young individuals with serious cardiac abnormalities may be identified if the significance of small QRS complexes is elucidated. The prevalence of small QRS complexes in the general population is 0.3-2% but there is paucity of data on prevalence and significance on small QRS complexes in young non-athletic individuals aged 17-35 years old. This study will allow the investigators to identify the prevalence and significance of small QRS complexes in athletes and non-athletes aged 17-35 years old potentially identifying young vulnerable individuals at risk of sudden cardiac death. These results should enable informed clinical decisions (at national and international level) following pre-participation screening evaluation and help ultimately to identify young individuals and athletes who are genuinely deemed to be at risk of sudden cardiac death (SCD) whilst providing appropriate reassurance to those with normal QRS voltages. This study will also potentially aid the investigators in updating the current recommendations on ECG interpretation in athletes which will influence future international ECG recommendations in athletes.This would be a cross-sectional observational study involving 240 participants aged 17-35 years old. This will involve 4 groups; 60 athletes with low QRS voltage and 60 age and sex matched control group of athletes with normal QRS voltage, 60 non-athletes with low QRS voltage and 60 age and sex matched controls with normal QRS voltage.

ELIGIBILITY:
Inclusion Criteria:

* No cardiovascular symptoms
* Body mass index <30.

Exclusion Criteria:

* Individuals with cardiac symptoms;
* Past medical history of cardiac disease, previous myocarditis or lung disease;
* Individuals with pacemakers or defibrillators
* Family history of SCD <40 years old or cardiomyopathy
* Pregnant women
* Advanced kidney and/or liver disease
* Known thyroid disease,
* T-wave inversion or other training unrelated ECG changes
* Known significant valvular heart disease or intra-cardiac shunt on echocardiography.

Ages: 17 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: 240 total study population:
  * 60 athletes with low QRS voltage and 60 age and sex matched control group of athletes with normal QRS voltage
  * 60 non-athletes with low QRS voltage and 60 age and sex matched controls with normal QRS voltage
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2023-10-09 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence of low QRS voltages in athletes and young non-athletic population on ECG analysis | 36 months
  Prevalence data will be obtained from existing ECG database of athletes and young people who have been screened by Cardiac risk in the young.
Prevalence of myocardial fibrosis in the young athletic and non-athletic population with low QRS | 36 months
  Participants satisfying inclusion criteria will undergo a cardiac MRI at a single time point to identify those with late gadolinium enhancement (indication of myocardial fibrosis)

SECONDARY OUTCOMES:
The proportion of individuals with low QRS complexes and myocardial fibrosis with rare protein altering variant in a cardiomyopathy gene. | 36 months
  A subgroup of athletes and young health individuals with low QRS voltages and myocardial fibrosis on cardiac MRI will undergo genetic analysis to identify the presence of protein altering genetic variants in known cardiomyopathy causing genes
The proportion of individuals with low QRS complexes and myocardial fibrosis with exercise related ventricular premature beats or a ventricular premature beat burden of > 500 beats on a Holter monitor | 36 months
  All participants will undergo cardiopulmonary exercise tests and 24 hour holter monitoring to identify presence of exercise related ventricular premature beats and a ventricular premature beat burden of > 500 beats on a Holter monitor

CONTACTS AND LOCATIONS:
Overall Officials: Sabiha Gati, MBBS, Principal Investigator — Royal Brompton & Harefield NHS Foundation Trust
Locations (1):
- Royal Brompton Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-06-22): https://cdn.clinicaltrials.gov/large-docs/33/NCT05799833/Prot_SAP_000.pdf
  • Informed Consent Form (2023-06-22): https://cdn.clinicaltrials.gov/large-docs/33/NCT05799833/ICF_001.pdf